CLINICAL TRIAL: NCT03878160
Title: Mindfulness-Based Cognitive Therapy Delivered Via Group Videoconferencing for Acute Coronary Syndrome Patients With Elevated Depression Symptoms
Brief Title: MBCT Delivered Via Group Videoconferencing for ACS Patients With Elevated Depression Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Christina Luberto, Clinical Psychology Fellow, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P001000; 1K23AT009715-01A1 (NIH)
Record Dates: First submitted 2019-02-26; First posted 2019-03-18 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Acute Coronary Syndrome; Depression; Myocardial Infarction; Unstable Angina; STEMI; NSTEMI - Non-ST Segment Elevation MI
Keywords: Mindfulness; Acute Coronary Syndrome; Videoconferencing; Depression
MeSH Terms: conditions — Acute Coronary Syndrome; Depression; Myocardial Infarction; Angina, Unstable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Approximately 20 individual interviews of ACS patients with elevated depression symptoms stratified by time since ACS (e.g. within the past 2 years or greater than 2 years ago), with 10 participants per strata. There will be approximately 10 individual interviews with ACS patients who are interested in treatment but not currently depressed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women and Men, <2 years, Individual Interview (Other): Individual interviews for women and men who have experienced an ACS within the past 2 years and have elevated depression symptoms.
  Interventions: Other: Individual Interview
- Women and Men, >2 years, Individual Interview (Other): Individual interviews for women and men who have experienced an ACS greater than 2 years ago and have elevated depression symptoms.
  Interventions: Other: Individual Interview
- Women and Men, Lifetime History of ACS, Individual Interview (Other): Individual interviews for women and men who have experienced an ACS at some point in their life and do not have elevated depression symptoms.
  Interventions: Other: Individual Interview

INTERVENTIONS:
Other: Individual Interview — Individual Interviews will focus on exploring (a) changes after ACS, such as psychosocial changes and health behavior changes; (b) specific preferences for the MBCT intervention; and (c) potential barriers and facilitators of group videoconferencing and (d) blood spot data collection. Individual interviews will use a semi-structured interview guide. Individual interviews will be conducted until thematic saturation is reached. Individual interviews will be audio-recorded for transcription and data analysis.

SUMMARY:
The objective of this study is to identify Acute Coronary Syndromes (ACS) patients' specific needs and preferences for depression treatment via in-person or virtual individual interviews to (a) guide MBCT adaptation; and identify barriers and facilitators to (b) group videoconferencing delivery, and (c) blood spot data collection to enhance feasibility. Through qualitative measures participants will report specific physical, cognitive, and behavioral symptoms to be targeted in the intervention, discuss barriers and facilitators to participating in a video-conference treatment program and completing blood spot data collection procedures.

DETAILED DESCRIPTION:
This is a qualitative research study that will involve individual interviews of ACS patients with elevated depression symptoms (stratified by time since ACS [≤2 years and >2 years post ACS]; N=10 participants per strata) to explore patients' treatment needs and preferences for an adapted MBCT intervention, and barriers and facilitators for future intervention research procedures (i.e., videoconferencing delivery of the intervention and collection of dried blood spots). It will also involve individual interviews of ACS patients without elevated depression symptoms (N=10) to better understand the needs of ACS patients who are interested in treatment but not currently depressed, in order to inform future outreach and treatment development efforts (total N=30). Interviews will be conducted either in person, by phone, or by video conference.

Participants will be recruited in several ways. First, participants will be identified using the MGH Research Patient Data Registry (RPDR). Participants will be pre-screened for eligibility and sent an opt-out letter. Patients will have the option to opt out via phone or email. Patients who do not opt out and meet eligibility requirements will be contacted via phone. Over the phone, patients who express interest in the study will complete an eligibility screen; patients who meet study eligibility criteria will then complete a verbal consent to enroll in the study. Second, patients will be recruited through advertisements (e.g., flyers, brochures) placed throughout inpatient and/or outpatient hospital clinics, community mental health clinics, community businesses (e.g. coffee shops) and social media platforms. The advertisements will ask patients to contact study staff if they are interested in learning more about the study, and the screening procedures will be the same as those described above for RPDR patients. Lastly, patients will be recruited via direct referrals from their providers (e.g., cardiologists, psychiatrists). We will inform providers about the study (e.g., via short presentations at their team meetings) and provide them with advertisement materials to give to their patients. The patients may either contact study staff directly using the information their provider gave them, and/or the provider will contact the study team with the patient's information so that the study team may reach out to the patient. Providers will obtain verbal permission from the patient for the research team to contact them.

Once enrolled, participants will partake in a semi-structured in-person individual interview. Individual interviews will be stratified by time since ACS and depressive symptoms and will explore (a) emotional symptoms; (b) health behavior challenges; (c) specific preferences for the MBCT intervention; and (d) potential barriers and facilitators of group videoconferencing and (e) blood spot data collection. Participants will also complete a survey detailing depression symptoms, trait mindfulness, health behaviors, and other psychological, behavioral, and physical constructs that may potentially be impacted by the MBCT intervention in subsequent trials will be measured. Data collected from the individual interviews will be used to guide MBCT adaptations and research procedures for future clinical trials.

ELIGIBILITY:
Inclusion criteria for depressed sample:

1. Lifetime ACS per medical record (for Partners' patients only) and/or patient confirmation
2. Current elevated depression symptoms (PHQ-9≥10)
3. Age 35-85 years
4. Access to high-speed internet

Exclusion criteria for depressed sample :

1. Active suicidal ideation or past-year psychiatric hospitalization
2. Non-English-speaking
3. Cognitive impairments preventing informed consent.

Inclusion criteria for non-depressed sample:

1. Lifetime ACS per medical record (for Partners' patients only) and/or patient confirmation
2. Age 35-85 years
3. Access to high-speed internet

Exclusion criteria for non-depressed sample:

1. Active suicidal ideation or past-year psychiatric hospitalization
2. Non-English-speaking
3. Cognitive impairments preventing informed consent.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Luberto, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spek V, Cuijpers P, Nyklicek I, Riper H, Keyzer J, Pop V. Internet-based cognitive behaviour therapy for symptoms of depression and anxiety: a meta-analysis. Psychol Med. 2007 Mar;37(3):319-28. doi: 10.1017/S0033291706008944. Epub 2006 Nov 20. PMID 17112400
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Kvedar J, Coye MJ, Everett W. Connected health: a review of technologies and strategies to improve patient care with telemedicine and telehealth. Health Aff (Millwood). 2014 Feb;33(2):194-9. doi: 10.1377/hlthaff.2013.0992. PMID 24493760
- [Background] Uchino BN. Social support and health: a review of physiological processes potentially underlying links to disease outcomes. J Behav Med. 2006 Aug;29(4):377-87. doi: 10.1007/s10865-006-9056-5. Epub 2006 Jun 7. PMID 16758315
- [Background] Uchino BN, Cacioppo JT, Kiecolt-Glaser JK. The relationship between social support and physiological processes: a review with emphasis on underlying mechanisms and implications for health. Psychol Bull. 1996 May;119(3):488-531. doi: 10.1037/0033-2909.119.3.488. PMID 8668748
- [Background] House JS, Landis KR, Umberson D. Social relationships and health. Science. 1988 Jul 29;241(4865):540-5. doi: 10.1126/science.3399889.
- [Background] Mohr DC, Burns MN, Schueller SM, Clarke G, Klinkman M. Behavioral intervention technologies: evidence review and recommendations for future research in mental health. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):332-8. doi: 10.1016/j.genhosppsych.2013.03.008. Epub 2013 May 8. PMID 23664503
- [Background] Ayala GX, Elder JP. Qualitative methods to ensure acceptability of behavioral and social interventions to the target population. J Public Health Dent. 2011 Winter;71 Suppl 1(0 1):S69-79. doi: 10.1111/j.1752-7325.2011.00241.x. PMID 21656958
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Miller G, Chen E, Cole SW. Health psychology: developing biologically plausible models linking the social world and physical health. Annu Rev Psychol. 2009;60:501-24. doi: 10.1146/annurev.psych.60.110707.163551. PMID 19035829
- [Background] Huffman JC, Celano CM, Beach SR, Motiwala SR, Januzzi JL. Depression and cardiac disease: epidemiology, mechanisms, and diagnosis. Cardiovasc Psychiatry Neurol. 2013;2013:695925. doi: 10.1155/2013/695925. Epub 2013 Apr 7. PMID 23653854
- [Background] Miller EM, McDade TW. A highly sensitive immunoassay for interleukin-6 in dried blood spots. Am J Hum Biol. 2012 Nov-Dec;24(6):863-5. doi: 10.1002/ajhb.22324. Epub 2012 Oct 5. PMID 23042671
- [Background] McDade TW, Williams S, Snodgrass JJ. What a drop can do: dried blood spots as a minimally invasive method for integrating biomarkers into population-based research. Demography. 2007 Nov;44(4):899-925. doi: 10.1353/dem.2007.0038. PMID 18232218
- [Background] Skogstrand K, Thorsen P, Norgaard-Pedersen B, Schendel DE, Sorensen LC, Hougaard DM. Simultaneous measurement of 25 inflammatory markers and neurotrophins in neonatal dried blood spots by immunoassay with xMAP technology. Clin Chem. 2005 Oct;51(10):1854-66. doi: 10.1373/clinchem.2005.052241. Epub 2005 Aug 4. PMID 16081507
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Background] Celano CM, Huffman JC. Depression and cardiac disease: a review. Cardiol Rev. 2011 May-Jun;19(3):130-42. doi: 10.1097/CRD.0b013e31820e8106. PMID 21464641
- [Background] van Melle JP, de Jonge P, Spijkerman TA, Tijssen JG, Ormel J, van Veldhuisen DJ, van den Brink RH, van den Berg MP. Prognostic association of depression following myocardial infarction with mortality and cardiovascular events: a meta-analysis. Psychosom Med. 2004 Nov-Dec;66(6):814-22. doi: 10.1097/01.psy.0000146294.82810.9c. PMID 15564344
- [Background] Lichtman JH, Bigger JT Jr, Blumenthal JA, Frasure-Smith N, Kaufmann PG, Lesperance F, Mark DB, Sheps DS, Taylor CB, Froelicher ES; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Epidemiology and Prevention; American Heart Association Interdisciplinary Council on Quality of Care and Outcomes Research; American Psychiatric Association. Depression and coronary heart disease: recommendations for screening, referral, and treatment: a science advisory from the American Heart Association Prevention Committee of the Council on Cardiovascular Nursing, Council on Clinical Cardiology, Council on Epidemiology and Prevention, and Interdisciplinary Council on Quality of Care and Outcomes Research: endorsed by the American Psychiatric Association. Circulation. 2008 Oct 21;118(17):1768-75. doi: 10.1161/CIRCULATIONAHA.108.190769. Epub 2008 Sep 29. PMID 18824640
- [Background] Huffman JC, Celano CM. Depression in cardiovascular disease: From awareness to action. Trends Cardiovasc Med. 2015 Oct;25(7):623-4. doi: 10.1016/j.tcm.2015.02.007. Epub 2015 Feb 20. No abstract available. PMID 25910599
- [Background] Dickens C, Cherrington A, Adeyemi I, Roughley K, Bower P, Garrett C, Bundy C, Coventry P. Characteristics of psychological interventions that improve depression in people with coronary heart disease: a systematic review and meta-regression. Psychosom Med. 2013 Feb;75(2):211-21. doi: 10.1097/PSY.0b013e31827ac009. Epub 2013 Jan 16. PMID 23324874
- [Background] Whalley B, Thompson DR, Taylor RS. Psychological interventions for coronary heart disease: cochrane systematic review and meta-analysis. Int J Behav Med. 2014 Feb;21(1):109-21. doi: 10.1007/s12529-012-9282-x. PMID 23179678
- [Background] Burg MM, Lesperance F, Rieckmann N, Clemow L, Skotzko C, Davidson KW. Treating persistent depressive symptoms in post-ACS patients: the project COPES phase-I randomized controlled trial. Contemp Clin Trials. 2008 Mar;29(2):231-40. doi: 10.1016/j.cct.2007.08.003. Epub 2007 Sep 5. PMID 17904917
- [Background] Segal ZV, Bieling P, Young T, MacQueen G, Cooke R, Martin L, Bloch R, Levitan RD. Antidepressant monotherapy vs sequential pharmacotherapy and mindfulness-based cognitive therapy, or placebo, for relapse prophylaxis in recurrent depression. Arch Gen Psychiatry. 2010 Dec;67(12):1256-64. doi: 10.1001/archgenpsychiatry.2010.168. PMID 21135325
- [Background] Kuyken W, Hayes R, Barrett B, Byng R, Dalgleish T, Kessler D, Lewis G, Watkins E, Brejcha C, Cardy J, Causley A, Cowderoy S, Evans A, Gradinger F, Kaur S, Lanham P, Morant N, Richards J, Shah P, Sutton H, Vicary R, Weaver A, Wilks J, Williams M, Taylor RS, Byford S. Effectiveness and cost-effectiveness of mindfulness-based cognitive therapy compared with maintenance antidepressant treatment in the prevention of depressive relapse or recurrence (PREVENT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):63-73. doi: 10.1016/S0140-6736(14)62222-4. Epub 2015 Apr 20. PMID 25907157
- [Background] Kuyken W, Byford S, Taylor RS, Watkins E, Holden E, White K, Barrett B, Byng R, Evans A, Mullan E, Teasdale JD. Mindfulness-based cognitive therapy to prevent relapse in recurrent depression. J Consult Clin Psychol. 2008 Dec;76(6):966-78. doi: 10.1037/a0013786. PMID 19045965
- [Background] Eisendrath SJ, Gillung E, Delucchi K, Mathalon DH, Yang TT, Satre DD, Rosser R, Sipe WE, Wolkowitz OM. A Preliminary Study: Efficacy of Mindfulness-Based Cognitive Therapy versus Sertraline as First-line Treatments for Major Depressive Disorder. Mindfulness (N Y). 2015 Jun 1;6(3):475-482. doi: 10.1007/s12671-014-0280-8. PMID 26085853
- [Background] Black DS, Slavich GM. Mindfulness meditation and the immune system: a systematic review of randomized controlled trials. Ann N Y Acad Sci. 2016 Jun;1373(1):13-24. doi: 10.1111/nyas.12998. Epub 2016 Jan 21. PMID 26799456
- [Background] Chambers R, Gullone E, Allen NB. Mindful emotion regulation: An integrative review. Clin Psychol Rev. 2009 Aug;29(6):560-72. doi: 10.1016/j.cpr.2009.06.005. Epub 2009 Jun 23. PMID 19632752
- [Background] Oikonomou MT, Arvanitis M, Sokolove RL. Mindfulness training for smoking cessation: A meta-analysis of randomized-controlled trials. J Health Psychol. 2017 Dec;22(14):1841-1850. doi: 10.1177/1359105316637667. Epub 2016 Apr 4. PMID 27044630
- [Background] Katterman SN, Kleinman BM, Hood MM, Nackers LM, Corsica JA. Mindfulness meditation as an intervention for binge eating, emotional eating, and weight loss: a systematic review. Eat Behav. 2014 Apr;15(2):197-204. doi: 10.1016/j.eatbeh.2014.01.005. Epub 2014 Feb 1. PMID 24854804
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Younge JO, Wery MF, Gotink RA, Utens EM, Michels M, Rizopoulos D, van Rossum EF, Hunink MG, Roos-Hesselink JW. Web-Based Mindfulness Intervention in Heart Disease: A Randomized Controlled Trial. PLoS One. 2015 Dec 7;10(12):e0143843. doi: 10.1371/journal.pone.0143843. eCollection 2015. PMID 26641099
- [Background] Boggs JM, Beck A, Felder JN, Dimidjian S, Metcalf CA, Segal ZV. Web-based intervention in mindfulness meditation for reducing residual depressive symptoms and relapse prophylaxis: a qualitative study. J Med Internet Res. 2014 Mar 24;16(3):e87. doi: 10.2196/jmir.3129. PMID 24662625
- [Background] Zernicke KA, Campbell TS, Speca M, McCabe-Ruff K, Flowers S, Carlson LE. A randomized wait-list controlled trial of feasibility and efficacy of an online mindfulness-based cancer recovery program: the eTherapy for cancer applying mindfulness trial. Psychosom Med. 2014 May;76(4):257-67. doi: 10.1097/PSY.0000000000000053. PMID 24804884
- [Background] Campo RA, Bluth K, Santacroce SJ, Knapik S, Tan J, Gold S, Philips K, Gaylord S, Asher GN. A mindful self-compassion videoconference intervention for nationally recruited posttreatment young adult cancer survivors: feasibility, acceptability, and psychosocial outcomes. Support Care Cancer. 2017 Jun;25(6):1759-1768. doi: 10.1007/s00520-017-3586-y. Epub 2017 Jan 19. PMID 28105523
- [Background] Wolever RQ, Bobinet KJ, McCabe K, Mackenzie ER, Fekete E, Kusnick CA, Baime M. Effective and viable mind-body stress reduction in the workplace: a randomized controlled trial. J Occup Health Psychol. 2012 Apr;17(2):246-258. doi: 10.1037/a0027278. Epub 2012 Feb 20. PMID 22352291
- [Background] Lichtman JH, Froelicher ES, Blumenthal JA, Carney RM, Doering LV, Frasure-Smith N, Freedland KE, Jaffe AS, Leifheit-Limson EC, Sheps DS, Vaccarino V, Wulsin L; American Heart Association Statistics Committee of the Council on Epidemiology and Prevention and the Council on Cardiovascular and Stroke Nursing. Depression as a risk factor for poor prognosis among patients with acute coronary syndrome: systematic review and recommendations: a scientific statement from the American Heart Association. Circulation. 2014 Mar 25;129(12):1350-69. doi: 10.1161/CIR.0000000000000019. Epub 2014 Feb 24. PMID 24566200
- [Background] Kaptein KI, de Jonge P, van den Brink RH, Korf J. Course of depressive symptoms after myocardial infarction and cardiac prognosis: a latent class analysis. Psychosom Med. 2006 Sep-Oct;68(5):662-8. doi: 10.1097/01.psy.0000233237.79085.57. Epub 2006 Sep 20. PMID 16987947
- [Background] Messay B, Lim A, Marsland AL. Current understanding of the bi-directional relationship of major depression with inflammation. Biol Mood Anxiety Disord. 2012 Feb 28;2:4. doi: 10.1186/2045-5380-2-4. PMID 22738397
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Ziegelstein RC, Fauerbach JA, Stevens SS, Romanelli J, Richter DP, Bush DE. Patients with depression are less likely to follow recommendations to reduce cardiac risk during recovery from a myocardial infarction. Arch Intern Med. 2000 Jun 26;160(12):1818-23. doi: 10.1001/archinte.160.12.1818. PMID 10871976
- [Background] Whooley MA, de Jonge P, Vittinghoff E, Otte C, Moos R, Carney RM, Ali S, Dowray S, Na B, Feldman MD, Schiller NB, Browner WS. Depressive symptoms, health behaviors, and risk of cardiovascular events in patients with coronary heart disease. JAMA. 2008 Nov 26;300(20):2379-88. doi: 10.1001/jama.2008.711. PMID 19033588
- [Background] Davidson KW, Rieckmann N, Clemow L, Schwartz JE, Shimbo D, Medina V, Albanese G, Kronish I, Hegel M, Burg MM. Enhanced depression care for patients with acute coronary syndrome and persistent depressive symptoms: coronary psychosocial evaluation studies randomized controlled trial. Arch Intern Med. 2010 Apr 12;170(7):600-8. doi: 10.1001/archinternmed.2010.29. PMID 20386003
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] Chu H, Yang J, Mi S, Bhuyan SS, Li J, Zhong L, Liu S, Tao Z, Li J, Chen H. Tumor necrosis factor-alpha G-308 A polymorphism and risk of coronary heart disease and myocardial infarction: A case-control study and meta-analysis. J Cardiovasc Dis Res. 2012 Apr;3(2):84-90. doi: 10.4103/0975-3583.95359. PMID 22629023
- [Background] Celano CM, Beale EE, Beach SR, Belcher AM, Suarez L, Motiwala SR, Gandhi PU, Gaggin H, Januzzi JL Jr, Healy BC, Huffman JC. Associations Between Psychological Constructs and Cardiac Biomarkers After Acute Coronary Syndrome. Psychosom Med. 2017 Apr;79(3):318-326. doi: 10.1097/PSY.0000000000000404. PMID 27749683
- [Background] Goldsmith DR, Rapaport MH, Miller BJ. A meta-analysis of blood cytokine network alterations in psychiatric patients: comparisons between schizophrenia, bipolar disorder and depression. Mol Psychiatry. 2016 Dec;21(12):1696-1709. doi: 10.1038/mp.2016.3. Epub 2016 Feb 23. PMID 26903267
- [Background] Hannestad J, DellaGioia N, Bloch M. The effect of antidepressant medication treatment on serum levels of inflammatory cytokines: a meta-analysis. Neuropsychopharmacology. 2011 Nov;36(12):2452-9. doi: 10.1038/npp.2011.132. Epub 2011 Jul 27. PMID 21796103
- [Background] Kappelmann N, Lewis G, Dantzer R, Jones PB, Khandaker GM. Antidepressant activity of anti-cytokine treatment: a systematic review and meta-analysis of clinical trials of chronic inflammatory conditions. Mol Psychiatry. 2018 Feb;23(2):335-343. doi: 10.1038/mp.2016.167. Epub 2016 Oct 18. PMID 27752078
- [Background] Raison CL, Capuron L, Miller AH. Cytokines sing the blues: inflammation and the pathogenesis of depression. Trends Immunol. 2006 Jan;27(1):24-31. doi: 10.1016/j.it.2005.11.006. Epub 2005 Nov 28. PMID 16316783
- [Background] Ridker PM, Rifai N, Pfeffer M, Sacks F, Lepage S, Braunwald E. Elevation of tumor necrosis factor-alpha and increased risk of recurrent coronary events after myocardial infarction. Circulation. 2000 May 9;101(18):2149-53. doi: 10.1161/01.cir.101.18.2149. PMID 10801754
- [Background] Finucane A, Mercer SW. An exploratory mixed methods study of the acceptability and effectiveness of Mindfulness-Based Cognitive Therapy for patients with active depression and anxiety in primary care. BMC Psychiatry. 2006 Apr 7;6:14. doi: 10.1186/1471-244X-6-14. PMID 16603060
- [Background] Chiesa A, Mandelli L, Serretti A. Mindfulness-based cognitive therapy versus psycho-education for patients with major depression who did not achieve remission following antidepressant treatment: a preliminary analysis. J Altern Complement Med. 2012 Aug;18(8):756-60. doi: 10.1089/acm.2011.0407. Epub 2012 Jul 13. PMID 22794787
- [Background] Levine GN, Lange RA, Bairey-Merz CN, Davidson RJ, Jamerson K, Mehta PK, Michos ED, Norris K, Ray IB, Saban KL, Shah T, Stein R, Smith SC Jr; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Hypertension. Meditation and Cardiovascular Risk Reduction: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2017 Sep 28;6(10):e002218. doi: 10.1161/JAHA.117.002218. PMID 28963100
- [Background] Fredrickson BL, Cohn MA, Coffey KA, Pek J, Finkel SM. Open hearts build lives: positive emotions, induced through loving-kindness meditation, build consequential personal resources. J Pers Soc Psychol. 2008 Nov;95(5):1045-1062. doi: 10.1037/a0013262. PMID 18954193
- [Background] Post SG. Altuism, happiness, and health: it's good to be good. Int J Behav Med. 2005;12(2):66-77. doi: 10.1207/s15327558ijbm1202_4. PMID 15901215
- [Background] Mookadam F, Arthur HM. Social support and its relationship to morbidity and mortality after acute myocardial infarction: systematic overview. Arch Intern Med. 2004 Jul 26;164(14):1514-8. doi: 10.1001/archinte.164.14.1514. PMID 15277281
- [Background] Schreier HM, Schonert-Reichl KA, Chen E. Effect of volunteering on risk factors for cardiovascular disease in adolescents: a randomized controlled trial. JAMA Pediatr. 2013 Apr;167(4):327-32. doi: 10.1001/jamapediatrics.2013.1100. PMID 23440253
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Background] Hofmann SG. Interpersonal Emotion Regulation Model of Mood and Anxiety Disorders. Cognit Ther Res. 2014 Oct;38(5):483-492. doi: 10.1007/s10608-014-9620-1. PMID 25267867
- [Background] Hibbard JH, Mahoney ER, Stock R, Tusler M. Do increases in patient activation result in improved self-management behaviors? Health Serv Res. 2007 Aug;42(4):1443-63. doi: 10.1111/j.1475-6773.2006.00669.x. PMID 17610432
- [Background] Brewer JA, Elwafi HM, Davis JH. Craving to quit: psychological models and neurobiological mechanisms of mindfulness training as treatment for addictions. Psychol Addict Behav. 2013 Jun;27(2):366-79. doi: 10.1037/a0028490. Epub 2012 May 28. PMID 22642859
- [Background] Vujanovic AA, Bonn-Miller MO, Bernstein A, McKee LG, Zvolensky MJ. Incremental validity of mindfulness skills in relation to emotional dysregulation among a young adult community sample. Cogn Behav Ther. 2010;39(3):203-13. doi: 10.1080/16506070903441630. PMID 20182933
- [Background] Hutcherson CA, Seppala EM, Gross JJ. Loving-kindness meditation increases social connectedness. Emotion. 2008 Oct;8(5):720-4. doi: 10.1037/a0013237. PMID 18837623
- [Background] Abbott RA, Whear R, Rodgers LR, Bethel A, Thompson Coon J, Kuyken W, Stein K, Dickens C. Effectiveness of mindfulness-based stress reduction and mindfulness based cognitive therapy in vascular disease: A systematic review and meta-analysis of randomised controlled trials. J Psychosom Res. 2014 May;76(5):341-51. doi: 10.1016/j.jpsychores.2014.02.012. Epub 2014 Mar 11. PMID 24745774
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Mohr DC, Ho J, Duffecy J, Baron KG, Lehman KA, Jin L, Reifler D. Perceived barriers to psychological treatments and their relationship to depression. J Clin Psychol. 2010 Apr;66(4):394-409. doi: 10.1002/jclp.20659. PMID 20127795
- [Background] Romano MF, Sardella MV, Alboni F. Web Health Monitoring Survey: A New Approach to Enhance the Effectiveness of Telemedicine Systems. JMIR Res Protoc. 2016 Jun 6;5(2):e101. doi: 10.2196/resprot.5187. PMID 27268949
- [Background] Mitzner TL, Boron JB, Fausset CB, Adams AE, Charness N, Czaja SJ, Dijkstra K, Fisk AD, Rogers WA, Sharit J. Older Adults Talk Technology: Technology Usage and Attitudes. Comput Human Behav. 2010 Nov 1;26(6):1710-1721. doi: 10.1016/j.chb.2010.06.020. PMID 20967133
- [Background] Botsis T, Hartvigsen G. Current status and future perspectives in telecare for elderly people suffering from chronic diseases. J Telemed Telecare. 2008;14(4):195-203. doi: 10.1258/jtt.2008.070905. PMID 18534954
- [Background] Mikolasek M, Berg J, Witt CM, Barth J. Effectiveness of Mindfulness- and Relaxation-Based eHealth Interventions for Patients with Medical Conditions: a Systematic Review and Synthesis. Int J Behav Med. 2018 Feb;25(1):1-16. doi: 10.1007/s12529-017-9679-7. PMID 28752414
- [Background] Gotink RA, Younge JO, Wery MF, Utens EMWJ, Michels M, Rizopoulos D, van Rossum LFC, Roos-Hesselink JW, Hunink MMG. Online mindfulness as a promising method to improve exercise capacity in heart disease: 12-month follow-up of a randomized controlled trial. PLoS One. 2017 May 9;12(5):e0175923. doi: 10.1371/journal.pone.0175923. eCollection 2017. PMID 28486559
- [Background] Wahbeh H, Goodrich E, Oken BS. Internet-based Mindfulness Meditation for Cognition and Mood in Older Adults: A Pilot Study. Altern Ther Health Med. 2016 Mar-Apr;22(2):44-53. PMID 27036056
- [Background] Luberto CM, White C, Sears RW, Cotton S. Integrative medicine for treating depression: an update on the latest evidence. Curr Psychiatry Rep. 2013 Sep;15(9):391. doi: 10.1007/s11920-013-0391-2. PMID 23943471
- [Background] Strawn JR, Cotton S, Luberto CM, Patino LR, Stahl LA, Weber WA, Eliassen JC, Sears R, DelBello MP. Neural Function Before and After Mindfulness-Based Cognitive Therapy in Anxious Adolescents at Risk for Developing Bipolar Disorder. J Child Adolesc Psychopharmacol. 2016 May;26(4):372-9. doi: 10.1089/cap.2015.0054. Epub 2016 Jan 19. PMID 26783833
- [Background] Kraemer KM, Luberto CM, O'Bryan EM, Mysinger E, Cotton S. Mind-Body Skills Training to Improve Distress Tolerance in Medical Students: A Pilot Study. Teach Learn Med. 2016;28(2):219-28. doi: 10.1080/10401334.2016.1146605. PMID 27064724
- [Background] Luberto CM, McLeish AC, Robertson SA, Avallone KM, Kraemer KM, Jeffries ER. The role of mindfulness skills in terms of distress tolerance: a pilot test among adult daily smokers. Am J Addict. 2014 Mar-Apr;23(2):184-8. doi: 10.1111/j.1521-0391.2013.12096.x. Epub 2013 Aug 31. PMID 25187054
- [Background] Huffman JC, Beach SR, Suarez L, Mastromauro CA, DuBois CM, Celano CM, Rollman BL, Januzzi JL. Design and baseline data from the Management of Sadness and Anxiety in Cardiology (MOSAIC) randomized controlled trial. Contemp Clin Trials. 2013 Nov;36(2):488-501. doi: 10.1016/j.cct.2013.09.012. Epub 2013 Oct 1. PMID 24090821
- [Background] Huffman JC, Mastromauro CA, Beach SR, Celano CM, DuBois CM, Healy BC, Suarez L, Rollman BL, Januzzi JL. Collaborative care for depression and anxiety disorders in patients with recent cardiac events: the Management of Sadness and Anxiety in Cardiology (MOSAIC) randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):927-35. doi: 10.1001/jamainternmed.2014.739. PMID 24733277
- [Background] Huffman JC, Mastromauro CA, Sowden G, Fricchione GL, Healy BC, Januzzi JL. Impact of a depression care management program for hospitalized cardiac patients. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):198-205. doi: 10.1161/CIRCOUTCOMES.110.959379. Epub 2011 Mar 8. PMID 21386067
- [Background] Park ER, Traeger L, Vranceanu AM, Scult M, Lerner JA, Benson H, Denninger J, Fricchione GL. The development of a patient-centered program based on the relaxation response: the Relaxation Response Resiliency Program (3RP). Psychosomatics. 2013 Mar-Apr;54(2):165-74. doi: 10.1016/j.psym.2012.09.001. Epub 2013 Jan 22. PMID 23352048
- [Background] Yeh GY, Wood MJ, Lorell BH, Stevenson LW, Eisenberg DM, Wayne PM, Goldberger AL, Davis RB, Phillips RS. Effects of tai chi mind-body movement therapy on functional status and exercise capacity in patients with chronic heart failure: a randomized controlled trial. Am J Med. 2004 Oct 15;117(8):541-8. doi: 10.1016/j.amjmed.2004.04.016. PMID 15465501
- [Background] Yeh GY, McCarthy EP, Wayne PM, Stevenson LW, Wood MJ, Forman D, Davis RB, Phillips RS. Tai chi exercise in patients with chronic heart failure: a randomized clinical trial. Arch Intern Med. 2011 Apr 25;171(8):750-7. doi: 10.1001/archinternmed.2011.150. PMID 21518942
- [Background] Yeh GY, Chan CW, Wayne PM, Conboy L. The Impact of Tai Chi Exercise on Self-Efficacy, Social Support, and Empowerment in Heart Failure: Insights from a Qualitative Sub-Study from a Randomized Controlled Trial. PLoS One. 2016 May 13;11(5):e0154678. doi: 10.1371/journal.pone.0154678. eCollection 2016. PMID 27177041
- [Background] Yeh GY, Wang C, Wayne PM, Phillips RS. The effect of tai chi exercise on blood pressure: a systematic review. Prev Cardiol. 2008 Spring;11(2):82-9. doi: 10.1111/j.1751-7141.2008.07565.x. PMID 18401235
- [Background] Yeh GY, Wang C, Wayne PM, Phillips R. Tai chi exercise for patients with cardiovascular conditions and risk factors: A SYSTEMATIC REVIEW. J Cardiopulm Rehabil Prev. 2009 May-Jun;29(3):152-60. doi: 10.1097/HCR.0b013e3181a33379. PMID 19471133
- [Background] Matchar DB, Jacobson A, Dolor R, Edson R, Uyeda L, Phibbs CS, Vertrees JE, Shih MC, Holodniy M, Lavori P; THINRS Executive Committee and Site Investigators. Effect of home testing of international normalized ratio on clinical events. N Engl J Med. 2010 Oct 21;363(17):1608-20. doi: 10.1056/NEJMoa1002617. PMID 20961244
- [Background] Siebenhofer A, Jeitler K, Horvath K, Habacher W, Schmidt L, Semlitsch T. Self-management of oral anticoagulation. Dtsch Arztebl Int. 2014 Feb 7;111(6):83-91. doi: 10.3238/arztebl.2014.0083. PMID 24622604
- [Background] Osler M, Martensson S, Wium-Andersen IK, Prescott E, Andersen PK, Jorgensen TS, Carlsen K, Wium-Andersen MK, Jorgensen MB. Depression After First Hospital Admission for Acute Coronary Syndrome: A Study of Time of Onset and Impact on Survival. Am J Epidemiol. 2016 Feb 1;183(3):218-26. doi: 10.1093/aje/kwv227. Epub 2016 Jan 5. PMID 26740025
- [Background] Carney RM, Freedland KE. Treatment-resistant depression and mortality after acute coronary syndrome. Am J Psychiatry. 2009 Apr;166(4):410-7. doi: 10.1176/appi.ajp.2008.08081239. Epub 2009 Mar 16. PMID 19289455
- [Background] Stafford L, Berk M, Jackson HJ. Validity of the Hospital Anxiety and Depression Scale and Patient Health Questionnaire-9 to screen for depression in patients with coronary artery disease. Gen Hosp Psychiatry. 2007 Sep-Oct;29(5):417-24. doi: 10.1016/j.genhosppsych.2007.06.005. PMID 17888808
- [Background] McManus D, Pipkin SS, Whooley MA. Screening for depression in patients with coronary heart disease (data from the Heart and Soul Study). Am J Cardiol. 2005 Oct 15;96(8):1076-81. doi: 10.1016/j.amjcard.2005.06.037. Epub 2005 Aug 30. PMID 16214441
- [Background] Thombs BD, de Jonge P, Coyne JC, Whooley MA, Frasure-Smith N, Mitchell AJ, Zuidersma M, Eze-Nliam C, Lima BB, Smith CG, Soderlund K, Ziegelstein RC. Depression screening and patient outcomes in cardiovascular care: a systematic review. JAMA. 2008 Nov 12;300(18):2161-71. doi: 10.1001/jama.2008.667. PMID 19001627
- [Background] Beach SR, Januzzi JL, Mastromauro CA, Healy BC, Beale EE, Celano CM, Huffman JC. Patient Health Questionnaire-9 score and adverse cardiac outcomes in patients hospitalized for acute cardiac disease. J Psychosom Res. 2013 Nov;75(5):409-13. doi: 10.1016/j.jpsychores.2013.08.001. Epub 2013 Aug 13. PMID 24182627
- [Background] Swenson JR, O'Connor CM, Barton D, Van Zyl LT, Swedberg K, Forman LM, Gaffney M, Glassman AH; Sertraline Antidepressant Heart Attack Randomized Trial (SADHART) Group. Influence of depression and effect of treatment with sertraline on quality of life after hospitalization for acute coronary syndrome. Am J Cardiol. 2003 Dec 1;92(11):1271-6. doi: 10.1016/j.amjcard.2003.08.006. PMID 14636902
- [Background] Bambauer KZ, Aupont O, Stone PH, Locke SE, Mullan MG, Colagiovanni J, McLaughlin TJ. The effect of a telephone counseling intervention on self-rated health of cardiac patients. Psychosom Med. 2005 Jul-Aug;67(4):539-45. doi: 10.1097/01.psy.0000171810.37958.61. PMID 16046365
- [Background] Mendes de Leon CF, Czajkowski SM, Freedland KE, Bang H, Powell LH, Wu C, Burg MM, DiLillo V, Ironson G, Krumholz HM, Mitchell P, Blumenthal JA; ENRICHD investigators. The effect of a psychosocial intervention and quality of life after acute myocardial infarction: the Enhancing Recovery in Coronary Heart Disease (ENRICHD) clinical trial. J Cardiopulm Rehabil. 2006 Jan-Feb;26(1):9-13; quiz 14-5. doi: 10.1097/00008483-200601000-00002. PMID 16617220
- [Background] Fung IN, Kim HL. Skin prick testing in patients using beta-blockers: a retrospective analysis. Allergy Asthma Clin Immunol. 2010 Jan 20;6(1):2. doi: 10.1186/1710-1492-6-2. PMID 20298514
- [Background] McDade TW, Leonard WR, Burhop J, Reyes-Garcia V, Vadez V, Huanca T, Godoy RA. Predictors of C-reactive protein in Tsimane' 2 to 15 year-olds in lowland Bolivia. Am J Phys Anthropol. 2005 Dec;128(4):906-13. doi: 10.1002/ajpa.20222. PMID 16118783
- [Background] McDade TW, Stallings JF, Worthman CM. Culture change and stress in Western Samoan youth: Methodological issues in the cross-cultural study of stress and immune function. Am J Hum Biol. 2000 Nov 1;12(6):792-802. doi: 10.1002/1520-6300(200011/12)12:63.0.CO;2-F. PMID 11534070
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Kistin C, Silverstein M. Pilot Studies: A Critical but Potentially Misused Component of Interventional Research. JAMA. 2015 Oct 20;314(15):1561-2. doi: 10.1001/jama.2015.10962. No abstract available. PMID 26501530
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Noone C, Hogan MJ. A randomised active-controlled trial to examine the effects of an online mindfulness intervention on executive control, critical thinking and key thinking dispositions in a university student sample. BMC Psychol. 2018 Apr 5;6(1):13. doi: 10.1186/s40359-018-0226-3. PMID 29622047
- [Background] Bowen S, Marlatt A. Surfing the urge: brief mindfulness-based intervention for college student smokers. Psychol Addict Behav. 2009 Dec;23(4):666-71. doi: 10.1037/a0017127. PMID 20025372
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186
- [Background] Nolen-Hoeksema S. Responses to depression and their effects on the duration of depressive episodes. J Abnorm Psychol. 1991 Nov;100(4):569-82. doi: 10.1037//0021-843x.100.4.569. PMID 1757671
- [Background] DiMatteo MR, Hays RD, Sherbourne CD. Adherence to cancer regimens: implications for treating the older patient. Oncology (Williston Park). 1992 Feb;6(2 Suppl):50-7. PMID 1532737
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- See also: Mindfulness-Based Cognitive Therapy Associated with Decreases in C - reactive protein in Major Depressive Disorder: A Pilot Study — https://www.researchgate.net/publication/317262864_Mindfulness-Based_Cognitive_Therapy_Associated_with_Decreases_in_C_-_reactive_protein_in_Major_Depressive_Disorder_A_Pilot_Study
- See also: A Systematic Review and Meta-analysis of the Effects of Meditation on Empathy, Compassion, and Prosocial Behaviors — https://www.researchgate.net/publication/320578887_A_Systematic_Review_and_Meta-analysis_of_the_Effects_of_Meditation_on_Empathy_Compassion_and_Prosocial_Behaviors
- See also: Mindfulness Interventions Delivered by Technology Without Facilitator Involvement: What Research Exists and What Are the Clinical Outcomes? — https://link.springer.com/article/10.1007/s12671-016-0548-2
- See also: Cognitive/affective and somatic/affective symptoms of depression in patients with heart disease and their association with cardiovascular prognosis: a meta-analysis — https://pdfs.semanticscholar.org/42c9/32a3c6d2a97407d7a34c342aee2fd2c39f04.pdf
- See also: Risk modification after myocardial infarction — https://www.researchgate.net/publication/19863972_Risk_modification_after_myocardial_infarction
- See also: Computer use by older adults: A multi-disciplinary review — http://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.458.1584&rep=rep1&type=pdf
- See also: Mindfulness Skills and Emotion Regulation: The Mediating Role of Coping Self-Efficacy — https://www.researchgate.net/publication/257795383_Mindfulness_Skills_and_Emotion_Regulation_The_Mediating_Role_of_Coping_Self-Efficacy
- See also: Mindfulness Skills and Emotion Regulation: the Mediating Role of Coping Self-Efficacy — https://www.infona.pl/resource/bwmeta1.element.springer-a4e1cb80-ca25-3231-9895-88757786f5b2
- See also: Breathing retraining for African-American adolescents with asthma: a pilot study of a school-based randomized controlled trial — https://search.pedro.org.au/search-results/record-detail/45938
- See also: Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale — https://link.springer.com/article/10.1023/B:JOBA.0000007455.08539.94
- See also: Measuring the Immeasurables: Development and Initial Validation of the Self-Other Four Immeasurables (SOFI) Scale Based on Buddhist Teachings on Loving Kindness, Compassion, Joy, and Equanimity — https://www.researchgate.net/publication/225563125_Measuring_the_Immeasurables_Development_and_Initial_Validation_of_the_Self-Other_Four_Immeasurables_SOFI_Scale_Based_on_Buddhist_Teachings_on_Loving_Kindness_Compassion_Joy_and_Equanimity
- See also: A Multidimensional Approach to Individual Differences in Empathy — https://www.uv.es/~friasnav/Davis_1980.pdf
- See also: Positive emotion dispositions differentially associated with Big Five personality and attachment style — https://asu.pure.elsevier.com/en/publications/positive-emotion-dispositions-differentially-associated-with-big-

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via the MGH Patient Hospital Data Registry, and provider referrals at an academic medical center between 02/2019-11/2019. The first participant was enrolled on 4/10/2019 and the last participant was enrolled on 11/11/2019.
Period: Overall Study
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Started | 7 | 9 | 11
Completed | 5 | 8 | 10
Not Completed | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Did not meet eligibility criteria, withdrawn by PI | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were healthy volunteers with a lifetime history of an acute coronary syndrome (ACS; e.g., MI, unstable angina).
Groups:
- Total: Total of all reporting groups
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview | Total
Number analyzed (Participants) | 5 | 8 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (12.7) | 64 (9.2) | 63.6 (6.0) | 63.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3
  Male | 5 | 5 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 8 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 5 | 6 | 9 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
PHQ-9 (Patient Health Questionnaire-9) Screen Score [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 (Patient Health Questionnaire-9) measures depressive symptoms, with scores ranging from 0-27, where lower scores indicate lesser depressive symptoms and higher scores indicate greater depressive symptoms. The units of the scale range from 0-3.
  units on a scale | 12.2 (3) | 12.3 (2.4) | 1.2 (1.3) | 7.4 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Changes After ACS
Description: This portion of the individual interview will focus on exploring changes experienced after an ACS, such as psychosocial changes and health behavior changes. Participants were individually interviewed via telephone using a semi-structured interview guide. Three independent coders conducted qualitative thematic analysis and results were analyzed within each group. The identified themes are reported, and the criteria used to determine the outcome measure is the number of participants who endorsed each theme.
Time Frame: one 30-90-minute session
Population: We explored the different types of changes patients might experience after ACS. We analyzed the data to identify the common themes regarding changes after ACS. We report the identified themes and the number of participants who expressed each theme.
Measure: Number; unit: participants
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 8 | 10
participants
  Positive health behavior changes | 3 | 3 | 10
  Adaptive perspectives | 1 | 0 | 5
  Emotional improvements | 0 | 1 | 1
  Social improvements | 1 | 0 | 5
  Activity limitations | 5 | 7 | 4
  Negative physical symptoms | 5 | 8 | 6
  Emotional problems | 3 | 8 | 6
  Social problems | 3 | 2 | 4
  Health behavior challenges | 2 | 5 | 0

2. Primary Outcome: Number of Participants With Perspectives on MBCT
Description: This portion of the individual interview will focus on exploring patients' perspectives toward an MBCT treatment approach. Participants were individually interviewed via telephone using a semi-structured interview guide. Three independent coders conducted qualitative thematic analysis and results were analyzed within each group. The identified themes are reported, and the criteria used to determine the outcome measure is the number of participants who endorsed each theme.
Time Frame: one 30-90-minute session
Population: We explored patients' willingness to participate in a group mindfulness program after ACS. We analyzed the data to identify the common themes. We report the identified themes and the number of participants who expressed each theme.
Measure: Number; unit: participants
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 8 | 10
participants
  Willing to get help | 3 | 8 | 8
  Willing to participate in a group program | 3 | 6 | 8
  Positive reaction to mindfulness | 4 | 7 | 7

3. Primary Outcome: Number of Participants With Perspectives on Videoconferencing
Description: This portion of the individual interview will focus on exploring perspectives regarding videoconferencing intervention delivery. Participants were individually interviewed via telephone using a semi-structured interview guide. Three independent coders conducted qualitative thematic analysis and results were analyzed within each group. Identified themes are reported, and the criteria used to determine the outcome measure is the number of participants upon interview who reported expressed each theme.
Time Frame: one 30-90-minute session
Population: We explored patients' perspectives toward using videoconferencing for a treatment program. We analyzed the data to identify the common themes regarding videoconferencing. We report the identified themes and the number of participants who expressed each theme.
Measure: Number; unit: participants
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 8 | 10
participants
  Willing to try videoconferencing | 3 | 7 | 8
  Logistical benefits | 5 | 5 | 7
  Social benefits | 2 | 1 | 1
  Technology limitations | 2 | 5 | 2
  Social limitations | 2 | 1 | 4

4. Primary Outcome: Number of Participants With Perspectives on Blood Spot Data Collection
Description: This portion of the individual interview will focus on exploring ACS patients who had perspectives on participating in a remote dried blood spot procedure. Participants were individually interviewed via telephone using a semi-structured interview guide. Three independent coders conducted qualitative thematic analysis and results were analyzed within each group. The criteria used to determine the outcome measure is the number of participants upon interview who reported any type of perspective on participating in a remote dried blood spot procedure (self-collection of dried blood spot via finger-prick). Please note that the number of perspectives reported for each theme can exceed the number of people per group because each participant reported multiple perspectives (e.g., both pros and cons of videoconferencing).
Time Frame: one 30-90-minute session
Population: We explored the patients' perspectives on completing a remote dried blood spot procedure. We analyzed the data to identify the common themes regarding this procedure. We report the identified themes and the number of participants who expressed each theme.
Measure: Number; unit: participants
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 8 | 10
participants
  Willing to complete DBS | 5 | 7 | 8
  Would need training | 2 | 5 | 2
  Would want more information about the rationale | 5 | 4 | 6

5. Secondary Outcome: Five Factor Mindfulness Questionnaire- 15 Item (FFMQ-15)
Description: This is a 15-item measure that measures mindfulness. This scale has five sub-scales: observing, describing, acting with awareness, accepting without judgment, and non-reactivity. The scoring scale ranges from 1, never or very rarely true to 5, very often or always true. Scale values range from 3-15 for each sub-scale, with higher values representing greater levels of individual mindfulness and lower values representing lowers levels of individual mindfulness. There is no total score for the measure; only individual sub-scales are reported. Data collection for this measurement is cross-sectional, and is collected during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: Participants were patients with a lifetime history of acute coronary syndrome (e.g., myocardial infarction, unstable angina).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 6 | 7
units on a scale
  Observing | 8 [7.5 to 10] | 9 [7 to 12] | 10 [8 to 14]
  Describing | 11 [8 to 13.5] | 9 [8 to 13] | 13 [11 to 14]
  Acting with awareness | 11 [8.5 to 13] | 9 [7 to 10] | 10 [9 to 14]
  Accepting without judgment | 11 [9.5 to 13.5] | 8 [6 to 10] | 14 [12 to 15]
  Nonreactivity | 11 [6.5 to 12.5] | 9.5 [7.75 to 10.5] | 14 [11 to 15]

6. Secondary Outcome: Perceived Stress Scale-4 (PSS-4)
Description: This is a 4-item scale that measures stress. The scoring scale ranges from 0,never, to 4, very often. The scale values range from 0-16 with higher values representing higher levels of individual stress and lower values representing lower levels of individual stress. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 7 | 7
units on a scale | 12 [11.5 to 14] | 14 [11 to 15] | 6 [4 to 8]

7. Secondary Outcome: Positive Affect Negative Affect Schedule (PANAS)
Description: This is a 20-question scale, composed of 2, 10-item scales that measure positive and negative affect. The scoring scale ranges from 1, very slightly or not at all, to 5, extremely. For this study, we will only use the positive affect sub-scale. The scale values for the positive affect sub-scale range from 10-50. Higher values on the positive affect scale represent higher levels of positive affect, whereas, lower values on the negative affect scale represent lower levels of positive affect. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 4 | 7 | 7
units on a scale | 22 [17.5 to 26.75] | 26 [21 to 32] | 34 [31 to 42]

8. Secondary Outcome: Rumination Response Scale (RRS)
Description: This is a 22-item scale that measures rumination. The scoring scale ranges from 1,almost never, to 4, almost always. The score values range from 22 to 88, where higher values represent higher levels of rumination and lower values represent lower levels of rumination. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 6 | 7
units on a scale | 41 [32 to 45.5] | 51.5 [33.75 to 56.25] | 31 [29 to 32]

9. Secondary Outcome: Self-Other Four Immeasurables (SOFI) Scale
Description: This is a 16-item scale that measures views toward the self and others. This measure consists of four sub-scales with four items each. The sub-scales measure positive views toward self, negative views toward self, positive views toward others, and negative views toward other. Only the positive-other sub-scale was used. The scoring scale ranges from 1, very slightly or not at all to 5, extremely, with sub-scale scores ranging from 4-20. Higher values represent higher levels of positive feelings toward others, and lower values represent lower levels of positive feelings toward others. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 4 | 6 | 7
units on a scale | 15 [12 to 15.75] | 12.5 [7.5 to 18.5] | 16 [15 to 18]

10. Secondary Outcome: Interpersonal Reactivity Index (IRI)
Description: This is a 14-item scale that measures empathy. The scoring scale ranges from 0, does not describe me well, to 4, describes me very well. The score values range from 0-56, where high values represent higher levels of empathy and lower values represent lower levels of empathy. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 4 | 7 | 6
units on a scale | 41 [36.25 to 45.75] | 39 [36 to 44] | 45 [35.25 to 51.25]

11. Secondary Outcome: Medical Outcomes Study - Specific Adherence Scale (MOS- SAS)
Description: This is a 3-item scale that measures health behaviors. The scoring scale ranges from 1, none of the time, to 6, all of the time. The scoring values range from 3-18, where higher values represent good health behavior and lower values represent poor health behavior. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 5 | 7 | 7
units on a scale | 11 [11 to 15.5] | 10 [10 to 12] | 13 [11 to 18]

12. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: This is a 9-item scale that measures depression. The scoring scale ranges from 0, not at all, to 3, nearly every day. The scoring values range from 0-18, where high values represent higher levels of depression and lower values represent lower levels of depression. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 4 | 6 | 6
units on a scale | 10.5 [8.25 to 12.75] | 16 [11.5 to 19.5] | 1.5 [0 to 4.5]

13. Secondary Outcome: Short-Form-12 (SF-12)
Description: This is a 12-item scale that measures health-related quality of life. The scoring scale from item 1 ranges from 1, excellent to 5, poor. The scoring scale for items 2 and 3 ranges from 1, limit you a lot to 3, not limit you at all. The scoring scale for questions 5-7 is represented by 1, yes or 2, no. The scoring scale for item 8 ranges from 1, not at all, to 5, extremely. The scoring scale for items 9-11 ranges from 1, all of the time, to 6, none of the time. The scoring scale for item 12 ranges from 1, all of the time to 5, none of the time. The total scoring values range from 12- 47, where higher values represent a higher quality of life and lower values represent a lower quality of life. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 3 | 7 | 7
units on a scale | 26 [25 to 25] | 22 [20 to 27] | 40 [33 to 42]

14. Secondary Outcome: Patient Reported Outcome Measurement Information System-Physical Function (PROMIS-29-PF)
Description: This is a 4-item scale that measures and evaluates physical health. The scoring scale ranges from 5, without any difficulty, to 1, unable to do. The scoring values range from 4-20, where high values represent good physical function and low values represent poor physical function. Data collection for this measurement is cross-sectional, and is performed during one, 30-90 minute time interval.
Time Frame: 30-90-minute study session
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
Number analyzed (Participants) | 3 | 7 | 7
units on a scale | 18 [13 to 13] | 12 [10 to 14] | 20 [13 to 20]

ADVERSE EVENTS:
Time Frame: 9 months
Description: No adverse events were reported as part of this study.
Arm/Group | Women and Men, <2 Years, Individual Interview | Women and Men, >2 Years, Individual Interview | Women and Men, Lifetime History of ACS, Individual Interview
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03878160/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT03878160/SAP_003.pdf